CLINICAL TRIAL: NCT04678349
Title: The Role of Partial Hydrolyzed Guar Gum in High Stoma Output Management Among Cancer Patients With Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: National Cancer Institute, Malaysia (Other Government)
Responsible Party: Principal Investigator, HO CHIOU YI, Principal Investigator, National Cancer Institute, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRR-19-3119-51323
Record Dates: First submitted 2020-11-24; First posted 2020-12-21 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHGG (Experimental): Patient who met inclusion criteria and consented during intervention period will be assigned as PHGG group. Surgical medical officer will obtain consent from eligible subject. After consented, subjects will be assessed weight and PG-SGA during admission. They will be given 4 scoops (40g) PHGG, which provide 160kcal, 0.24g protein, 30.4g soluble fibre, 40g carbohydrate and 0g sugar once allowed orally. Staff nurse in charged will monitor compliance of subject on the PHGG. Daily stoma output & consistency will be recorded and daily energy protein intake will be assessed by dietitian in charged. Renal profile will be taken daily as routine procedure for patients with ileostomy.
  Interventions: Dietary Supplement: PHGG
- CG (Other): Historical records of patients with ileostomy under conventional care from January 2016 to June 2019 (before started on PHGG) will be assessed and traced retrospectively from the medical system. Data will be recorded in data collection sheet.
  Interventions: Other: conventional care

INTERVENTIONS:
Dietary Supplement: PHGG — Subjects will be given 4 scoops (40g) PHGG, which provide 160kcal, 0.24g protein, 30.4g soluble fibre, 40g carbohydrate and 0g sugar, once allowed orally.
  Arms: PHGG
Other: conventional care — follow low fibre diet and anti-diarrhea drugs
  Arms: CG

SUMMARY:
this is a cross sectional intervention study to investigate the role of partial hydrolyzed guar gum in high stoma output management among cancer patients with ileostomy. This study hypotheses there is improvement in stoma output in PHGG if compare with control. There are two groups of subjects in this study. Conventional group (CG) will include retrospective historical data (those subjects with post-operative ileostomy) from Jan 2016 to June 2019. Intervention group (PHGG) will be subjects with ileostomy which involves prospective intervention by giving partial hydrolyzed guar gum upon start orally. Data on stoma output (volume & consistency), length of hospital stay, readmission within 30-days discharged and dietary intake will be recorded in data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with ileostomy
* At least 18 years of age
* Malaysian

Exclusion Criteria:

* Not cancer patients with ileostomy
* Patients who participate in other study at the same time
* Vulnerable subjects
* Palliative patients
* Patient has fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
ileostomy stoma output | up to 1 month
  consistency (bristrol stool chart; range 1-7; 1 hard while 7 watery)
ileostomy stoma output | up to 1 month
  volume (ml)

SECONDARY OUTCOMES:
Length of hospital stay | up to 1 month
  days of hospital stays
Readmission within 30-days discharged | up to 1 month
  readmit to ward due to complications after discharge
Dietary intake | up to 1 month
  energy (kcal/day)
dietary intake | up to 1 month
  protein intake (g/day)

CONTACTS AND LOCATIONS:
Overall Officials: ChiouYi Ho, Principal Investigator — Department of Dietetics and Food Service, Institut Kanser Negara
Locations (1):
- National Cancer Institute, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided